CLINICAL TRIAL: NCT04333563
Title: Non-invasive Neurally Adjusted Ventilator Assist or Continuous Positive Airway Pressure in Preterm Infants: A Randomized Crossover Study
Brief Title: Non-invasive Neurally Adjusted Ventilator Assist or Continuous Positive Airway Pressure in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 58386
Record Dates: First submitted 2020-04-01; First posted 2020-04-03 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-07

CONDITIONS: Premature Birth; Respiratory Distress Syndrome, Newborn
Keywords: Infants, preterm; Respiration, Artificial; Diaphragm; Intensive Care Units, Neonatal; Continuous Positive Airway Pressure; Non invasive neurally adjusted ventilator assist
MeSH Terms: conditions — Premature Birth; Respiratory Distress Syndrome, Newborn; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPAP (Active Comparator): respiratory stressed infants getting Continuous positive airway pressure (CPAP)
  Interventions: Device: CPAP; Device: NIV NAVA
- respiratory stressed infants getting NIV NAVA (Experimental): respiratory stressed infants getting Non-invasive neurally adjusted ventilatory assist (NIV NAVA)
  Interventions: Device: CPAP; Device: NIV NAVA

INTERVENTIONS:
Device: CPAP — Continuous positive airway pressure
Device: NIV NAVA — Non-invasive neurally adjusted ventilatory assist

SUMMARY:
Strategies to prevent lung injury, facilitate lung development, and to support the preterm infant's capacity to breathe are decisive. Continuous positive airway pressure (CPAP) is the gold standard in non-invasive breathing support in preterm infants with a positive pressure that keeps the alveoli slightly inflated during expiration. Non-invasive neurally adjusted ventilator assist (NIV NAVA) is a novel method of breathing support and uses the electrical activity from the diaphragm to trigger the ventilator and synchronize with the breathing cycle. During NIV NAVA the preterm infant controls the onset of the inspiration, the respiratory rate, inspiratory time and peak pressure. This method has the potential to improve the positive pressure transmission to the infant's lower airways, accurate synchronization with the breathing pattern and be a comfortable breathing support system for the preterm infant.

The investigators will compare the effect on breathing effort in preterm infants during continuous positive airway pressure and non-invasive neurally adjusted ventilatory assist measured by electrical activity in the diaphragm, respiratory vital signs, systematic clinical scoring of breathing effort and comfort, and parent reported outcomes.

DETAILED DESCRIPTION:
This is a randomized cross-over study with AB/BA sequences. The infants will receive both interventions in 4 hours intervals, a 30 minutes period to change the breathing support and a 30 minutes wash out period between interventions. Initially positive end expiratory pressure are set to 5 cm H2O and can be adjusted up to 7 cm H2O if needed decided by the medical team for both interventions. The neurally adjusted level will be set to obtain average Edi peak < 15 microvolt. Back-up setting and apnea time in the ventilator assist intervention (NIV NAVA) will be individualized according to clinical parameters in each preterm infant.

Modification approved by ethical committee REK 2021, 6th of August:

After two hours in each intervention, the nurse responsible for the infant will perform the clinical scoring. In addition it will be investigated if there is a difference in respiratory vital signs during skin to skin care and in the incubator. During each intervention period, the preterm infants are placed on the parent's chest skin to skin for at least one hour.

A modified version of the scoring tool will be used, i.e. without the item of nasal flaring and expiratory grunting. The headgear for CPAP and NIV NAVA covers parts of the nose and makes nasal flaring difficult to observe.

ELIGIBILITY:
Inclusion Criteria:

* spontaneously breathing preterm infants 24 to 96 hours old
* gestational age (GA) between week 28+0 and 31+6
* preterm infants with GA < 28+0 with a postmenstrual age (PMA) > 28 weeks
* at least 72 hours old treated with CPAP or NIV NAVA

Exclusion Criteria:

* preterm infants with severe congenital malformation
* need for vasopressors
* preterm children in need of a specific respiratory support system due to medical reasons

Ages: 24 Hours to 96 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2020-04-14 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Electrical activity of the diaphragm | 9 hours and 30 minutes
  Electromyography signals from the diaphragm in 30 second intervals

SECONDARY OUTCOMES:
Silverman Andersen Respiratory Severity Score | Three minutes
  The scoring tool consists of 5 categories and respiratory distress are graded from zero to two for each category. Respiratory distress gets worse the higher the total score gets.
Scoring blinded for the intervention | Three minutes video-recording
  During each intervention, the infants will be video recorded for a blinded assessment.
COMFORTneo pain scale | Three minutes
  Measuring pain and discomfort in a seven category scale graded from 1 - 5, where one is best and five is worse.
Parents opinion about the outcomes | Three minutes
  Three questions about their opinion about the interventions in a 5 point Likert scale
Respiratory rate | 30 second intervals
  Standard monitoring on IntelliVue monitor
Heart rate | 30 second intervals
  Standard monitoring on IntelliVue monitor
Oxygen saturation | 30 second intervals
  Standard monitoring on IntelliVue monitor
number of apneic episodes ≥ 20 seconds | 9 hours and 30 seconds
  Using trend function on the IntelliVue monitor

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Selvaag, md, Study Director — St Olavs Hospital, Barne- og ungdomsklinikk
Locations (1):
- Department of Pediatrics St Olavs Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Yes
Study protocol Statistical analysis Informed consent form
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 2022 and to 2027
URL: https://hilde.brenne@stolav.no